CLINICAL TRIAL: NCT01022372
Title: The Evaluation of Endometrial Biopsy in the Diagnosis of Endometriosis and Endometrioma: a Double Blind Study
Brief Title: Endometrial Biopsy as Diagnostic Method for Endometriosis and Endometrioma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Alaa S.MAHMOUD, SELCUK UNIVERSITY- MERAM MEDICAL FACULTY
Other Study IDs: 2009035
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2010-07

CONDITIONS: Women in the Reproductive Age Group; Undergoing Laparoscopy for Pelvic Pain and/or Infertility; Not Currently Receiving Hormonal Treatment for at Least 3 Months Prior to Laparoscopy.

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- control group
  Interventions: Procedure: Endometrial biopsy
- endometriosis group
  Interventions: Procedure: Endometrial biopsy
- endometrioma group
  Interventions: Procedure: Endometrial biopsy

INTERVENTIONS:
Procedure: Endometrial biopsy — For all the groups

SUMMARY:
Our aim was to evaluate the efficacy of examining endometrial biopsy specimens for nerve fibers as a diagnostic test for endometriosis and endometrioma in a double-blind comparison with diagnostic laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Women in the reproductive age group undergoing laparoscopy for pelvic pain and/or infertility, and not currently receiving hormonal treatment for at least 3 months prior to laparoscopy will be included in the study

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: women in the reproductive age group undergoing laparoscopy for pelvic pain and/or infertility, and not currently receiving hormonal treatment for at least 3 months prior to laparoscopy will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The density of nerve fibers in the endometrial biopsy sample. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The hospital of Meram medical Faculty, Konya, Turkey (Türkiye)